CLINICAL TRIAL: NCT02411019
Title: A Prospective, Observational, Open-label, Multi-center, Follow-up Clinical Study to Determine Recurrence of Cervical Intraepithelial Neoplasia and Evaluate the Long-term Safety of GX-188E, a DNA-based Therapeutic Vaccine, Administered Intramuscularly by Electroporation (EP) in Subjects Who Were Diagnosed With HPV(Human Papillomavirus) 16 or 18 Positive Cervical Intraepithelial Neoplasia 3 (CIN 3) and Participated in Phase 2 Trial (GX-188E_CIN3_P2)
Brief Title: Safety and Efficacy of GX-188E DNA Therapeutic Vaccine Administered by Electroporation After Observation
Acronym: GX-188E
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GX-188E_CIN3_P2_FU
Record Dates: First submitted 2015-03-16; First posted 2015-04-08 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Cervical Intraepithelial Neoplasia 3
Keywords: Phase 2 follow up; Cervical Intraepithelial Neoplasia; Adult; Safety; Efficacy
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — GX-188 vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and PBMC (peripheral blood mononeuclear cell)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational group: Subjects in the period less than 24 weeks after the final administration of GX-188E
  Interventions: Biological: GX-188E

INTERVENTIONS:
Biological: GX-188E — In phase II study, 72 patients were assigned to two dose groups (1mg and 4mg) and were administered three times with GX-188E by electroporation during an entire period of study. After the final administration, the follow-up will be conducted to investigate safety and efficacy aspects.
  Other Names: GX-188E administered by electrophoration

SUMMARY:
This study is to follow up on the change of immune response by measuring HPV type 16/18 E6 and E7 specific T cell response and lesion condition in subjects who have administered in DNA-based therapeutic vaccine.

DETAILED DESCRIPTION:
This is a follow-up study to investigate the change of immunogenicity and lesion condition in subjects with cervical intraepithelial neoplasia (CIN) 3 who have enrolled and participated GX-188E phase II trial(GX-188E_CIN3_P2).

Subjects will make visits 7 times for about three years from the last visit of GX-188E phase 2 trial (GX-188E_CIN3_P2).

The endpoints are to evaluate the change of immune response, involved lesion and infection status compared to that of the final visit in phase 2 trial (GX-188E_CIN3_P2).

ELIGIBILITY:
Inclusion Criteria:

* Those who voluntarily signed informed consent form
* The subjects who have participated in phase II trial(GX-188E_CIN3_P2)

Exclusion Criteria:

* The subjects who didn't receive GX-188E DNA vaccine during Phase II trial (GX-188E_CIN3_P2)
* The subjects, it is difficult to participate in this study continuously
* Any other ineligible condition at the discretion of the investigator that would be ineligible to participate the study

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The subjects who have completed the DNA vaccine administration of each dosage (1 and 4 mg).
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Safety assessment examined by physical examination, vital signs, ECG, clinical laboratory test etc | at week -18 and 130
  long term safety assessment of GX-188E DNA vaccine of subjects participated in GX-188E_ CIN3_P2 clinical trial
  - Safety profile would be examined by physical examination, vital signs, ECG, clinical laboratory test etc
lesion recurrence | at week -18 and 130
  The change of the CIN lesion (included cervical cancer) would be compared to that of the last visit in phase II study

SECONDARY OUTCOMES:
The change of HPV infection status | at week -18 and 130
  The change of HPV infection status would be compared to that of the last visit in phase II study.
The change of cytology test result | at week -18 and 130
  The change of cytology status would be compared to that of the last visit in phase II study.
The change of the immune response | at week -18 and 130
  It would be determined by evaluating HPV type 16/18 E6 and E7 specific T cell response (IFN-γ ELISPOT: enzyme-linked immunospot assay) using PBMC(peripheral blood monocyte).
Flt-3L(fms-related tyrosine kinase 3 ligand) concentration (Flt-3L ELISA) using plasma. | at week -18 and 130
  Pharmacodynamics evaluation of GX-188E
Survey of pregnancy and delivery | at week -18 and 130
  The matters relevant to the subject of pregnancy and delivery would be collected by survey to identify occurence, frequency and characteristic.

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Sup Park, M.D., Principal Investigator — The Catholic University of Korea; Tae-Jin Kim, M.D., Principal Investigator — Cheil General Hospital & Women's Healthcare Center; Jae-Kwan Lee, M.D., Principal Investigator — Korea University Guro Hospital; Chi-Heum Cho, M.D., Principal Investigator — Keimyung University Dongsan Medical Center
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea